CLINICAL TRIAL: NCT05324670
Title: Intervention Based on Didactic Model for Suicidal Behavior in the Framework of Impulsivity and Ideations.
Brief Title: Title: "Intervention Based on Didactic Model for Suicidal Behavior in the Framework of Impulsivity and Ideations."
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Islamic University, Islamabad (Other)
Responsible Party: Principal Investigator, Mudassar Abdullah, Mudassar Abdullah, International Islamic University, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSSSP
Record Dates: First submitted 2022-04-03; First posted 2022-04-12 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Suicidal Ideation and Behavior; Impulsivity
MeSH Terms: conditions — Suicidal Ideation; Behavior; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: Research design of the study will consists single-blind cluster randomized controlled trial (c-RCT). While Randomized Control Trial (RCT) will consists of two groups: written knowledge with explanation (experimental group) and written knowledge without explanation (control group).
Who Masked: Participant
Masking Description: Single blind Cluster randomized controlled trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental condition (Experimental): Didactic intervention based on religious teachings and cultural milieu, the experimental group will receive 12 sessions for three months, 4 sessions per month including focused group discussion.
  Interventions: Other: Didactic model for suicidal behavior in the framework of impulsivity and ideations
- Control condition (Other): They will have sessions like the experimental group but the control group will get the knowledge in the form of written material without any explanation (Information Leaflet).
  Interventions: Other: Didactic model for suicidal behavior in the framework of impulsivity and ideations

INTERVENTIONS:
Other: Didactic model for suicidal behavior in the framework of impulsivity and ideations — It will be in the form of lectures (Educational approach). Content will be developed one day before the commencement of the session. The Knowledge provided in the form of written material with proper explanation shall not exceed 30 minutes and a Focused group Discussion will be held at the end of each month.
  Other Names: Prophylactic Strategy Known as Didactic intervention

SUMMARY:
Suicide has become a major public health problem among young people around the world. This study will examine the effects of higher secondary school-based suicide prevention (HSSSP) program on youth suicidal thoughts and impulsive behavior (STIB). Therefore, the purpose of this study is to examine the effects of didactic approach for youth STIB on the HSSSP program.

This study is designed to address this issue at the secondary school level. Therefore, this research is divided into two studies. In the first study, our goal was to arrange a Baseline assessment for the screening process of adolescents at risk of suicide. while in second study we aim to implement a didactic approach based on religious teachings and culture milieu and examine its effects as an evidence based suicide prevention program.

DETAILED DESCRIPTION:
Suicide has become a major public health problem around the world. according to a recent report by the World Health Organization (WHO) suicide is the fourth leading cause of death among youth. Suicidal thoughts and suicide attempts are on the rise among youth. Therefore, evidence-based prevention programs need to fill this gap with interventions at the higher secondary schools.

For decades, research and prevention efforts have been failed in developing meaningful predictions and reductions in suicide. However, significant efforts are needed to stop the rising tide of suicide. For the purpose, it is important to understand the suicidal thought at first as not everyone who commits suicide attempts suicide first.

Therefore, in this study an attempt has been made to investigate profoundly the understanding of suicide which has been emerged a serious problem around the globe and in particular in Pakistani society. The researcher has planned to conduct psychological measures with established psychometric properties to look at the relationship between suicidal ideation and impulsivity anticipating suicidal behavior. During study the role of moderators i.e. social effectiveness and level of religiosity shall also be investigated. Findings of this study shall comprehensively provide data in order to design an inclusive prophylactic strategy known as didactic intervention to prevent the suicidal act before it occurs. It is expected that this approach grounded on religious teaching and cultural milieu in line with the best practices, will be adapted. Subsequently, this study also aims to evaluate the effectiveness of the didactic approach as an evidence based suicide prevention program in higher secondary schools with selective prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* Higher Secondary School Students
* Young people at risk of suicide: those who are impulsive and have suicidal thoughts.

Exclusion Criteria:

* Who has a history of suicide attempts

Ages: 12 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Barratt Impulsiveness scale | Assessment at baseline (after screening), 8th week after baseline (2 months), 16th week after baseline (4 months). The purpose of the outcome measure is to estimate the change from baseline assessment to follow-up.
  This is a 4-point likert scale and is scored in the following way; Rarely/Never= 1, Occasionally= 2, Often= 3 & Almost/Always= 4. It contains 30 items that describe common impulsive or non-impulsive behaviors and preferences.
Beck Scale for Suicidal Ideation | Assessment at baseline (after screening), 8th week after baseline (2 months), 16th week after baseline (4 months). The purpose of the outcome measure is to estimate the change from baseline assessment to follow-up.
  This scale entails of 19 items and measures 3 responses from Least severe= 0 to Most severe= 2

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS) | Assessment at baseline (after screening), 8th week after baseline (2 months), 16th week after baseline (4 months). The purpose of the outcome measure is to estimate the change from baseline assessment to follow-up.
  This scale consists of a set of three self-reported measures in the form of 4-point Likert severity/frequency format. Each scale contains 14 items, subdivided into 2-5 item subscales containing the same contents.
Stroop Test | Assessment at baseline (after screening), 8th week after baseline (2 months), 16th week after baseline (4 months). The purpose of the outcome measure is to estimate the change from baseline assessment to follow-up.
  The Stroop Color Test assesses the ability to prevent cognitive interference, which occurs while processing the stimulus feature affects the simultaneous processing of another attribute of the same stimulus.
Self-Efficacy scale | Assessment at baseline (after screening), 8th week after baseline (2 months), 16th week after baseline (4 months). The purpose of the outcome measure is to estimate the change from baseline assessment to follow-up.
  It is a 4-point Likert-type scale consisting of 10 items, and measures are taken in response from strongly disagree to strongly agree.
Religious commitment inventory (RCI-10) | Assessment at baseline (after screening), 8th week after baseline (2 months), 16th week after baseline (4 months). The purpose of the outcome measure is to estimate the change from baseline assessment to follow-up.
  This scale consists of 10 items. The responses are made in a 5 - point Likert format from Not at all to Totally true of me.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad T Khalily, Study Chair — Department of Psychology, IIUI
Locations (1):
- International Islamic University, Islamabad, Islamabad (CapitalTerritory), Pakistan

REFERENCES:
- [Result] Eggert LL, Thompson EA, Herting JR, Nicholas LJ. Reducing suicide potential among high-risk youth: tests of a school-based prevention program. Suicide Life Threat Behav. 1995 Summer;25(2):276-96. PMID 7570788
- [Result] Aseltine RH Jr, DeMartino R. An outcome evaluation of the SOS Suicide Prevention Program. Am J Public Health. 2004 Mar;94(3):446-51. doi: 10.2105/ajph.94.3.446. PMID 14998812
- [Result] Randell BP, Eggert LL, Pike KC. Immediate post intervention effects of two brief youth suicide prevention interventions. Suicide Life Threat Behav. 2001 Spring;31(1):41-61. doi: 10.1521/suli.31.1.41.21308. PMID 11326768